CLINICAL TRIAL: NCT05915585
Title: Efficacy of High-Intensity Laser Therapy for the Management of Eosinophilic Fasciitis: A Case Report
Brief Title: High-Intensity Laser Therapy for Eosinophilic Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010/012023
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Eosinophilic Fasciitis
MeSH Terms: conditions — Eosinophilic Fasciitis

STUDY DESIGN:
Intervention Model Description: Single participant case study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-Intensity Laser Therapy (HILT) (Experimental)
  Interventions: Device: High-Intensity Laser Therapy

INTERVENTIONS:
Device: High-Intensity Laser Therapy — The patient will receive HILT using the Mectronic Exand MY high-intensity laser system with the following parameters:
  Wavelength: 1064 nm (near-infrared) Power: 12 W Energy density: 8 J/cm² Pulse duration: 200 µs Treatment duration: 10 minutes Frequency: 3 sessions per week for 4 weeks Total energy delivered: 96 J per treatment session

SUMMARY:
Eosinophilic fasciitis (EF) is a rare musculoskeletal disorder characterized by inflammation and thickening of the fascia, leading to pain, stiffness, and functional impairment. Conventional treatment options include immunosuppressive medications, corticosteroids, and physical therapy. This case report will describe use of high-intensity laser therapy (HILT) using the Mectronic Exand MY high-intensity laser system in a patient with EF, highlighting its potential as an alternative or adjunct treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Eosinophilic fasciitis.

Exclusion Criteria:

* a diagnosis unrelated to Eosinophilic fasciitis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2023-06-18 (Estimated); Primary Completion 2023-07-19 (Estimated); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
Pain intensity via Numeric pain rating scale | Changes in pain intensity at baseline and 4 weeks
Functional outcomes via Disabilities of the Arm, Shoulder and Hand questionnaire (DASH) | Changes in DASH at baseline and 4 weeks
Quality of life via Short Form-36 Health Survey | Changes in Short Form-36 Health Survey at baseline and 4 weeks
Adverse event | 4 Weeks
  adverse events are recorded by the patient and therapist

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No